CLINICAL TRIAL: NCT05021731
Title: Comparison of 3-month Once-weekly Isoniazid Plus Rifapentine, 4-month Daily Rifampicin, and 3-month Daily Isoniazid Plus Rifampicin for the Treatment Latent Tuberculosis in Patients With End-stage Kidney Disease: A Randomised Clinical Trial
Brief Title: Short-course Rifamycin-based Regimens for Latent Tuberculosis in Patients With End-stage Kidney Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Miguel Santín (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Miguel Santín, Senior consultant in infectious diseases, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI21/00444
Record Dates: First submitted 2021-08-13; First posted 2021-08-25 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Latent Tuberculosis; Kidney Failure
Keywords: Tuberculosis; Rifamycins; Rifampicin; Rifapentine; Kidney failure
MeSH Terms: conditions — Latent Tuberculosis; Renal Insufficiency; Tuberculosis | interventions — Rifampin; Isoniazid; rifapentine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 3-month Isoniazid plus Rifampicin (Active Comparator): Daily isoniazid 300 mg plus rifampicin 600 mg for three months
  Interventions: Drug: Rifampicin plus Isoniazid
- 3-month Isoniazid plus Rifapentine (Experimental): Weekly isoniazid 900 mg plus rifapentine 900 mg for 12 weeks
  Interventions: Drug: Rifapentine plus Isoniazid
- 4-month Rifampicin (Experimental): Daily rifampicin 600 mg for four months
  Interventions: Drug: Rifampicin alone

INTERVENTIONS:
Drug: Rifampicin plus Isoniazid — Administration of rifampicin plus isoniazid for latent tuberculosis
  Arms: 3-month Isoniazid plus Rifampicin
Drug: Rifapentine plus Isoniazid — Administration of rifapentine plus isoniazid for latent tuberculosis
  Arms: 3-month Isoniazid plus Rifapentine
Drug: Rifampicin alone — Administration of rifampicin alone for latent tuberculosis
  Arms: 4-month Rifampicin

SUMMARY:
Objective To determine if treatment completion with a 4-month rifampin (4R) or 3-month rifapentine (P) + isoniazid (H) weekly for 12 weeks (3HP) regimens is better than with a 3-month (3HR) regimen for treatment of latent tuberculosis (TB) infection (LTBI) in patients with end stage kidney disease.

Methods Design: Multicenter, prospective, parallel-group, open-label, controlled clinical trial.

Study population: All adult patients with ESKD in who treatment for LTBI is prescribed at 7 hospitals.

Interventions: Patients who accept participation, will be randomly assigned to one of the 3 arms: 3HR (control) (90 doses), 4R (120 doses) or 3HP (12 doses).

Outcome: Proportion of participants who discontinue permanently the assigned treatment. Follow-up: Periodic assessment for permanent or temporary discontinuation, and adverse events of the assigned treatment.

Sample size: 225 subjects (75 per arm) will be needed to demonstrate, if exists, a 0.16 decrease in permanent discontinuation rates in the experimental arms (4R and 3HP) with respect to the control arm (3HR), with α= 0.025, β= 0.20, and 5% expected losses, and assuming a 0.25 proportion of permanent discontinuation in the control.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Stage 5 kidney disease (glomerular filtrate rate <15 mL/minute or under substitutive renal therapy
3. Informed written consent

Exclusion Criteria:

1. Prior allergy/intolerance to rifamycins or isoniazid
2. Pregnancy or breastfeeding
3. Pre-treatment transaminases (ALT and/or AST) >5-fold of normality titer
4. Concomitant drugs contraindicated with rifamycins
5. Having received rifamycins or isoniazid within the two previous weeks
6. Weigh <32 Kgs
7. Inability to understand the nature of the study or to give written consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Treatment completion | From date of randomization until the date of completion of the assigned treatment, or date of lost to follow-up, or date of death, whichever came first, assessed up to 16 weeks for the 3HR arm, 14 weeks for the 3HP arm, and 20 weeks for the 4R arm.
  Proportion of participants who complete the treatment assigned at randomization, defined as: 1) 90 doses within a maximum of 16 weeks, without interruptions longer than 2 weeks, and no more than in 2 occasions, for 3HR (control arm); 2) 12 doses within a maximum of 14 weeks, without interruptions longer than 10 days, for 3HP (experimental arm 1), and 3) 120 doses within a maximum of 20 weeks, without interruptions longer than 2 weeks, and no more than in two occasions, for 4R (experimental arm 2).

SECONDARY OUTCOMES:
Permanent discontinuation because of adverse events | From date of randomization until the date of completion of the assigned treatment, or date of lost to follow-up, or date of death, whichever came first, assessed up to 16 weeks for the 3HR arm, 14 weeks for the 3HP arm, and 20 weeks for the 4R arm.
  Proportion of participants who permanently discontinue the treatment assigned, because of adverse events, regardless the relationship of the event/s to the study treatment.
  Permanent discontinuation defined as: 1) not completion of 90 doses within a maximum of 16 weeks, without interruptions longer than 2 weeks, and no more than in 2 occasions, for 3HR (control arm); 2) not completion 12 doses within a maximum of 14 weeks, without interruptions longer than 10 days, for 3HP (experimental arm 1), and 3) not completion of 120 doses within a maximum of 20 weeks, without interruptions longer than 2 weeks, and no more than in two occasions, for 4R (experimental arm 2).
Permanent discontinuation because of adverse events related to the treatment | From date of randomization until the date of completion of the assigned treatment, or date of lost to follow-up, or date of death, whichever came first, assessed up to 16 weeks for the 3HR arm, 14 weeks for the 3HP arm, and 20 weeks for the 4R arm.
  Proportion of participants who permanently discontinue the treatment assigned, because of adverse events related to he study treatment
  Permanent discontinuation defined as: 1) not completion of 90 doses within a maximum of 16 weeks, without interruptions longer than 2 weeks, and no more than in 2 occasions, for 3HR (control arm); 2) not completion 12 doses within a maximum of 14 weeks, without interruptions longer than 10 days, for 3HP (experimental arm 1), and 3) not completion of 120 doses within a maximum of 20 weeks, without interruptions longer than 2 weeks, and no more than in two occasions, for 4R (experimental arm 2).
Death | From date of randomization until four weeks after completing the assigned treatment, or lost to follow-up, assessed up to 17 weeks for the 3HR arm, 15 weeks for the 3HP arm, and 21 weeks for the 4R arm.
  Number of participants who die while on the study, regardless of its relationship to the treatment assigned at randomization

REFERENCES:
- [Derived] Santin M, Perez-Recio S, Grijota MD, Anibarro L, Barcala JM, De Souza-Galvao ML, Gijon P, Luque R, Sanchez F; RIFAKiD team trial. Comparison of three short-course rifamycin-based regimens for the prevention of tuberculosis in patients with end-stage kidney disease: Study protocol for a randomised clinical trial (RIFAKiD-TB trial). PLoS One. 2022 Oct 21;17(10):e0276387. doi: 10.1371/journal.pone.0276387. eCollection 2022. PMID 36269714